CLINICAL TRIAL: NCT02519933
Title: A Comparison of Modified Non-transposed Brachiobasilic Arteriovenous Fistula and Brachiocephalic Arteriovenous Fistula in Hemodialysis Patients
Brief Title: A Comparison of mNT-BBAVF and BCAVF in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, Director of the department of Nephrology, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai10
Record Dates: First submitted 2015-07-21; First posted 2015-08-11 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Vascular Fistula
Keywords: hemodialysis; vascular access
MeSH Terms: conditions — Vascular Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mNT-BBAVF (Active Comparator): Patients in Chronic Kidney Disease (CKD) stage 4-5 without previous dysfunctional fistula access
  Interventions: Procedure: mNT-BBAVF
- BCAVF (Active Comparator): Patients in CKD stage 4-5 without previous dysfunctional fistula access
  Interventions: Procedure: BCAVF

INTERVENTIONS:
Procedure: mNT-BBAVF — mNT-BBAVF was performed under local anesthesia. A transverse incision of approximately 4 cm was made in the antecubital area. The basilic vein was isolated, and its side branches were ligated; followed by the isolation of brachial artery. A venotomy of 5 mm was performed, followed an arteriotomy of 5 mm. The two vessels then had a side-to-side anastomosis, followed by the ligation of the vein above anastomosis. All the perforating veins located in an area 2-4 cm down the antecubital fossa from anastomosis were separated and ligated carefully. After surgeries, all patients will be followed up for 12 months. The outcomes are patency (primary unassisted patency and secondary), complications and hemodynamic parameters (diameters, blood velocities and blood volume) detected by Ultrasound.
  Arms: mNT-BBAVF
Procedure: BCAVF — BCAVF was performed under local anesthesia. A transverse incision of approximately 4 cm in length was made in the medial antecubital area. The cephalic vein was isolated, followed by the isolation of brachial artery. The distal end of cephalic vein was ligated and dissected. Patency of the proximal vein was verified by the warmed saline injection. The artery was then incised after clamping, and an end-to-side anastomosis (4-0 silk suture) between the cephalic vein and the brachial artery was performed. At last the skin is sutured (1-0 silk suture). At last the skin is sutured. After surgeries, all patients will be followed up for 12 months. The outcomes are patency (primary unassisted patency and secondary), complications and hemodynamic parameters detected by Ultrasound.
  Arms: BCAVF

SUMMARY:
A well-functioning vascular access is essential for effective hemodialysis. The native arteriovenous fistula (AVF) is the preferred vascular access because of the lower thrombosis and infection risks compared to either synthetic arteriovenous grafts or central venous catheters. Brachiocephalic arteriovenous fistula (BCAVF) and transposed brachiobasilic arteriovenous fistula (T-BBAVF) are recommended when there is either a primary failure or no suitable vessels for the forearm fistula. However, BCAVF is frequently cannulated at the antecubital fossa, the risks of stenosis and thrombosis are high, which will compromise proper BCAVF function and survival. T-BBAVF is not only technically challenging, but also associates with severe arm swelling and pain. Thus, the investigators introduced a novel modified Non-transposed brachiobasilic arteriovenous fistula (mNT-BBAVF) for long-term hemodialysis patients. To confirm its efficacy, a prospective clinical study would be carried out.

DETAILED DESCRIPTION:
The study aims to compare the outcomes of a novel modified Non-transposed brachiobasilic arteriovenous fistula (mNT-BBAVF) and the standard brachiocephalic arteriovenous fistula (BCAVF) for long-term hemodialysis patients. Briefly, in mNT-BBAVF, a side-to-side anastomosis between the brachial artery and non-transposed proximal basilic vein is disposed, followed by the ligation of the vein above anastomosis. All the perforating in the surgical field should be ligated. All patients will be followed up for 12 months after surgeries. The outcomes includes: hemodynamic parameters (vessels's diameters, blood flow velocities and blood volumes) detected by ultrasound in 12 months, Complications in 1-month and 12-month, primary patency and secondary patency (cumulative patency).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years;
* Radial artery diameter <2.0 mm or cephalic vein diameter in the forearm <2.5 mm;
* Brachial artery diameter ≥ 2 mm

Exclusion Criteria:

* Stenosis or thrombosis present in the draining vein;
* A history of peripheral ischemia in upper extremities;
* Active local or systemic infections;
* Inability to consent for the procedure;
* Patients with previous dysfunctional forearm fistula.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04; Primary Completion 2018-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Primary unassited patency | 12 months
  The interval from the time of access creation to any first intervention (endovascular or surgical) designed to maintain or reestablish patency, access thrombosis.

SECONDARY OUTCOMES:
Cumulative patency | 12 month
  The interval from the time of access placement to access abandonment, including intervening (all surgical and endovascular interventions) designed to reestablish the functionality of thrombosed access.
Short-term complications | 1 month
  Complications of both mNT-BBAVF and BCAVF groups within 1 month (thrombosis, failure of maturation, bleeding, steal syndrome, arm edema and severe arm pain)
Long-term complications | 12 months
  Complications of both mNT-BBAVF and BCAVF groups within 12 months (thrombosis, stenosis and aneurysm).
Calculated blood flow volumes of the corresponding fistula segments | 12 months
  Blood flow volume (ml/min) = mean velocity (cm/s) * area (r2π) * 60 seconds.
Diameters of the veins and arteries in the corresponding arm | 12 months
  Vessels's diameters (cm) of the relevant veins (proximal cephalic vein, distal cephalic vein, distal basilic vein) and arteries (Subclavian artery, axillary artery, brachial artery, radial artery and ulnar artery) in the corresponding arm.
Blood flow velocities of the veins and arteries in the corresponding arm. | 12 months
  Blood flow velocities (cm/s) of the relevant veins (proximal cephalic vein, distal cephalic vein, distal basilic vein) and arteries (Subclavian artery, axillary artery, brachial artery, radial artery and ulnar artery) in the corresponding arm.

CONTACTS AND LOCATIONS:
Overall Officials: AI Peng, M.D., Ph.D., Principal Investigator — The Division of Nephrology & Rheumatology, Shanghai 10th People's Hospital
Locations (2):
- Rhode Island Hospital/Brown University Medicine School, Providence, Rhode Island, United States
- The Division of Nephrology & Rheumatology, Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No